CLINICAL TRIAL: NCT07199179
Title: Link Between Reduction of Suicide Ideation by Esketamine in Add-On and Initial Levels of Psychological Pain and Anhedonia
Acronym: IODA
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL24_0018
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Depression - Major Depressive Disorder; Depression Disorder; Suicide
Keywords: ESKETAMINE
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is looking at how intranasal esketamine (a nasal spray) can help reduce suicidal thoughts in patients with severe depression who are experiencing suicidal thoughts. Suicidal depression is a type of depression where people have active thoughts of suicide, which can be harder to treat with regular antidepressants. In fact, some people continue to have suicidal thoughts even after taking antidepressants.

Esketamine has already shown promise in helping reduce suicidal thoughts quickly-often within 24 hours-and these effects can last for up to 25 days. Researchers believe esketamine may work by improving mood-related symptoms like loss of pleasure (called anhedonia) and feelings of hopelessness, which are linked to suicidal thinking. They also think that psychological pain, or emotional distress, might play a role in how well esketamine helps reduce suicidal thoughts.

The goal of this study is to better understand how esketamine works to improve suicidal thoughts and whether certain factors (like mood symptoms or emotional pain) can predict which patients will benefit the most from this treatment.

This study uses data from two earlier clinical trials, called ASPIRE I (NCT03039192) and ASPIRE II (NCT03097133), that tested intranasal esketamine in patients with depression and suicidal thoughts. All data from these studies are publicly available and can be accessed and analyzed through the YODA (Yale University Open Data Access) platform, a database of clinical trial data that is accessible to external researchers.

ELIGIBILITY:
Inclusion Criteria:

* patients who participated in the ASPIRE I (NCT03039192) and ASPIRE II (NCT03097133)

Exclusion Criteria:

* Not applicable

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population includes the 456 patients enrolled in the ASPIRE I and ASPIRE II studies.
Sampling Method: Non-Probability Sample
Enrollment: 456 (Actual)
Dates: Start 2024-11-24 (Actual); Primary Completion 2025-11-24 (Estimated); Study Completion 2025-11-24 (Estimated)

PRIMARY OUTCOMES:
Anhedonia | Measured at 24 hours, 7 days, and 25 days after the first administration of intranasal esketamine vs. placebo
  The primary outcome measure is the level of anhedonia, assessed by items 5, 7, 8, and 10 of the Montgomery-Åsberg Depression Rating Scale (MADRS). These items evaluate the loss of interest or pleasure in usual activities, a key symptom related to both depression and suicidal ideation.
  A higher score indicates greater anhedonia, meaning a more severe loss of interest or pleasure. A decrease in the score over time suggests improvement in the patient's ability to experience pleasure.

SECONDARY OUTCOMES:
Psychological Pain | Measured at 24 hours, 7 days, and 25 days after the first administration of intranasal esketamine vs. placebo.
  Psychological pain assessed using specific items from the Suicide Ideation and Behavior Assessment Tool (SIBAT). The SIBAT includes items from both modules 2 and 3 that describe various dimensions of psychological pain.
  A higher score on the SIBAT indicates greater psychological pain, including emotional distress tied to suicidal ideation. A decrease in score suggests a reduction in psychological pain
Hopelessness | Measured at 24 hours, 7 days, and 25 days after the first administration of intranasal esketamine vs. placebo.
  Hopelessness is measured using the Beck Hopelessness Scale (BHS), which consists of 20 true/false items evaluating the patient's perception of hopelessness and their outlook on the future. A higher score indicates greater hopelessness. A decrease in the score indicates improvement in the patient's outlook and reduction in hopelessness.
Severity of Suicidal Thoughts | Measured at 24 hours, 7 days, and 25 days after the first administration of intranasal esketamine vs. placebo.
  Suicidal thoughts are assessed by a specific item on the Montgomery-Åsberg Depression Rating Scale (MADRS), which directly addresses the presence and severity of suicidal thoughts.
  Higher score indicates more severe suicidal thoughts.
  Suicidal severity is also assessed by The Clinical Global Impression-Severity Scale-Revised (CGI-SS-r). The scale evaluates both the presence and severity of suicidal thoughts and behaviors.
  higher score indicates more severe suicidal ideation
Frequency of Suicidal Ideation | Measured at 24 hours, 7 days, and 25 days after the first administration of intranasal esketamine vs. placebo.
  - Patient Reported : The frequency of suicidal ideation is reported by the patient using the Suicide Ideation and Behavior Assessment Tool (SIBAT). This assesses how often the patient experiences suicidal thoughts throughout the study period.
  A higher score indicates more frequent suicidal thoughts
  - Clinician Reported : The clinician evaluates the frequency of suicidal ideation based on observations using the Suicide Ideation and Behavior Assessment Tool (SIBAT). A higher score indicates more frequent suicidal ideation observed by the clinician
Depressive Symptoms Severity | Assessed at 24 hours, 7 days, and 25 days after the first administration of intranasal esketamine vs. placebo.
  Depressive symptoms are evaluated using the Montgomery-Åsberg Depression Rating Scale (MADRS), which includes 10 items assessing the severity of depression, including mood, anxiety, and cognitive symptoms.
  A higher score indicates more severe depressive symptoms (0-6: No depression or very mild depression, 7-20: Mild to moderate depression, 21-34: Moderate to severe depression, 35+: Severe depression).

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No